CLINICAL TRIAL: NCT06508866
Title: Timing And Typology of ConducTIon disturbanCes During TAVI: the TACTIC-TAVI Registry
Brief Title: Timing And Typology of ConducTIon disturbanCes During TAVI
Acronym: TACTIC-TAVI
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 3328
Record Dates: First submitted 2024-07-15; First posted 2024-07-18 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Aortic Stenosis, Severe
Keywords: TAVI; Pacemaker; aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The TACTIC-TAVI registry aims to collect information about a consecutive cohort of patients undergoing transcatheter aortic valve insertion. The registry is international, multi-centre and observational. The registry is planned to continue until the calculated sample size is achieved.

DETAILED DESCRIPTION:
All patients since February 2023 treated successfully with TAVI until the study endpoint will be deemed suitable for inclusion in the registry. The registry will:

1. collect the baseline clinical features of the study population.
2. evaluate the electrocardiogram (ECG) and contrast tomography (CT) scan parameters.
3. collect procedural characteristics including type and timing of any conduction disturbance
4. collect follow-up data including post-procedural ECG, echocardiographic and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients successfully undergoing transcatheter aortic valve implantation for native severe aortic stenosis.

-

Exclusion Criteria:

1. Presence of previously implanted permanent cardiac pacemaker.
2. Valve-in-valve procedures.
3. No pre-procedural electrocardiogram is available.
4. No pre-procedural contrast CT TAVI is available.
5. Enrollment in another clinical trial.
6. Patients aged less than 18 years old.
7. Patients who do not consent for their data to be included in the registry.
8. Failed transcatheter aortic valve deployment. -

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study is a retrospective and prospective registry aiming to observe intra-procedural conduction disturbances in patients undergoing TAVI for severe aortic stenosis. Patients will have no alteration to standard post-procedural management and will their have usual follow-up. There are four key time points: 1) pre-procedure 2) intra-procedure 3) post-procedure 4) discharge. The electrocardiogram will be assessed at timepoints 1-3 and requirement for permanent pacemaker insertion by timepoint 4.
Sampling Method: Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prediction of new requirement for permanent pacemaker after TAVI | 0-24 months
  The primary focus of the registry is evaluating which patient characteristics and conduction disturbances may help to predict the new requirement for permanent pacemaker after TAVI.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Mangieri, MD, Principal Investigator — Humanitas Research Horspital
Locations (1):
- IRCCS Istituo Clinico Humanitas, Rozzano, Milano, Italy